CLINICAL TRIAL: NCT00090662
Title: Collection of Data and Samples From Healthy Donors for Use in Translational Research
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040266; 04-I-0266
Record Dates: First submitted 2004-09-01; First posted 2004-09-02 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-05-15

CONDITIONS: Healthy Volunteer
Keywords: Cerebrospinal Fluid; Stool; Urine; Natural History; Skin; Sputum; Healthy Volunteer; HV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteer: Healthy volunteer

SUMMARY:
Increased numbers of white blood cells called eosinophils can cause disease. To investigate this disease, researchers need blood, urine, sputum, stool, cerebrospinal fluid, skin and/or bone marrow samples to compare to samples from patients with this problem. Some of the samples will be used for genetic testing or future research.

This study will last for about 10 years and will include a maximum of 50 paid volunteers ages 18 to 65.

DETAILED DESCRIPTION:
This protocol is designed to provide data and samples from paid volunteers for use in translational studies of eosinophilia and parasitic diseases. Donors meeting standard normal donor eligibility criteria will be recruited to undergo research procedures (infrared thermography and/or esophageal string test) and/or to donate blood, body fluid and/or tissue samples obtained using conventional techniques. The investigational nature of the studies in which their data and/or samples will be used, as well as the risks and benefits of the procedures, will be explained to all volunteers, and a signed informed consent document will be obtained. Volunteers will be compensated according to an established schedule based on the duration and discomfort of the donation. Samples provided through this protocol will be used solely for in vitro research and will be assigned a unique product number. The study investigators listed on this protocol will serve as the custodians of the code that links the product with a donor s identity. The nature of the in vitro studies in which the data and specimens collected in this study will be used is not the subject of this protocol and will be described in general terms only, since it involves several IRB-approved LPD protocols. Because some of these protocols require normal controls without a history of asthma or allergic disease, all subjects will undergo a standardized allergy/asthma history at enrollment. Serum immunoglobulin levels and a basic RAST panel may be performed on sera from some normal donors, and some normal donors may be asked to undergo pulmonary function testing.

ELIGIBILITY:
* Eligibility criteria for volunteer whole blood donation are based on the Standards of the AABB(2) and the Code of Federal Regulation 21 CFR 640(3). Specific criteria follow:

INCLUSION CRITERIA (blood, urine, stool, infrared thermograpy, photography, gastrointestinal secretion, pulmonary function testing

and/or sputum donation)

* ability to sign informed consent
* healthy male or female
* 18-85 years of age

EXCLUSION CRITERIA (blood, urine, stool, infrared thermograpy, photography, gastrointestinal secretion, pulmonary function testing

and/or sputum donation)

* pregnancy
* weight <110 pounds
* history of heart, lung, kidney disease, chronic anemia or bleeding disorders

Eligibility for tissue biopsy donation (other than skin) will be determined by the protocol under which the procedure is performed and the physician performing the procedure.

Eligibility criteria for volunteer bone marrow, skin and cerebrospinal fluid donation are more stringent than those for other specimen donations to minimize risk of procedure complications and maximize utility of specimens for study:

INCLUSION CRITERIA (bone marrow, cerebrospinal fluid and/or skin donation)

* ability to sign informed consent
* healthy, male or female
* 18-65 years of age
* willingness to provide concurrent blood sample

EXCLUSION CRITERIA (bone marrow, cerebrospinal fluid and/or skin donation)

* a known bleeding disorder, low platelets (<100k) or taking medications that interfere with blood clotting, such as aspirin, non-steroidal anti-inflammatory agents or warfarin
* anemia (hemoglobin less than 12.3 mg/dL)
* evidence of an immune deficiency, such as HIV infection or cancer
* pregnancy
* taking a medication that affects the immune response within the past month, including oral, intravenous, or injectable steroids
* allergic to xylocaine
* have taken an investigational drug in the last 6 months
* any other medical condition that the investigator feels puts the participant at too high a risk for participation

  * warfarin and/or heparin treatment will not be stopped so that a subject can participate in this protocol. If warfarin or heparin was recently discontinued, a subject can be enrolled, but no bone marrow procedures will be performed until the PT is < 15.5 seconds and the PTT is within normal range. For other agents that interfere with blood clotting without prolonging the PT, a 7- day washout period will be required before bone marrow sampling, skin biopsy or lumbar puncture.

Additional exclusion criteria (cerebrospinal fluid)

-Previous diagnosis of central nervous system pathology (including tumors,

inflammatory conditions, infection, seizure disorder, spina bifida)

* History of spinal surgery with hardware placement
* History of any spinal surgery or injections of the lumbosacral spine
* Headache on the day of donation

Additional exclusion criteria (skin biopsy)

-History of keloid or abnormal scar formation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2004-12-09 (Actual)

PRIMARY OUTCOMES:
- To provide an IRB-approved mechanism for the collection of peripheral blood, urine, sputum, stool, cerebrospinal fluid, skin biopsy and bone marrow samples from paid, volunteer donors for use in in vitro studies. | 50 years
  - To provide adequate and complete informed consent to the donors of research blood samples, and to assure that the education, counseling and protection of the study subjects from research risks is performed in accordance with IRB, OHRP, and other applicable Federal regulatory standards.

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Klion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No.

REFERENCES:
- [Derived] Bennuru S, Kodua F, Drame PM, Dahlstrom E, Nutman TB. A Novel, Highly Sensitive Nucleic Acid Amplification Test Assay for the Diagnosis of Loiasis and its Use for Detection of Circulating Cell-Free DNA. J Infect Dis. 2023 Oct 3;228(7):936-943. doi: 10.1093/infdis/jiad186. PMID 37243712
- [Derived] Stokes K, Yoon P, Makiya M, Gebreegziabher M, Holland-Thomas N, Ware J, Wetzler L, Khoury P, Klion AD. Mechanisms of glucocorticoid resistance in hypereosinophilic syndromes. Clin Exp Allergy. 2019 Dec;49(12):1598-1604. doi: 10.1111/cea.13509. Epub 2019 Oct 27. PMID 31657082
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-I-0266.html